CLINICAL TRIAL: NCT06918925
Title: A Double-blind, Placebo-controlled, First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single- and Multiple-ascending Doses of JUV-161 Administered Subcutaneously to Healthy Adult Volunteers.
Brief Title: First-In-Human Study to Evaluate Single and Multiple Ascending Doses of JUV-161 in Healthy Adult Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Juvena Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JUV-161-101
Record Dates: First submitted 2025-03-24; First posted 2025-04-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Intervention Model Description: double-blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JUV-161 (Active Comparator): Single-ascending dose administration of JUV-161/ 5 cohorts of 6 subjects SAD 1 JUV-161 0.10 mg/kg 6 subjects SAD 2 JUV-161 0.30 mg/kg 6 subjects SAD 3 JUV-161 1.00 mg/kg 6 subjects SAD 4 JUV-161 3.00 mg/kg 6 subjects SAD 5 JUV-161 5.0 mg/kg 6 subjects SAD 6 JUV-161 10.0mg/kg 6 subjects
  MAD 1 JUV-161 0.10 mg/kg 6 subjects X 3 doses MAD2 JUV-161 3.00 mg/kg 6 subjects X 3 doses MAD3 JUV-161 5.0 mg/kg 6 subjects x 3 doses
  Interventions: Drug: JUV-161, Placebo
- Placebo-Controlled (Placebo Comparator): SAD1 placebo 2 subjects X 1 dose SAD 2 placebo 2 subjects X 1 dose SAD 3 placebo 2 subjects X 1 dose SAD 4 placebo 2 subjects X 1 dose SAD 5 placebo 2 subjects X 1 dose SAD 6 placebo 2 subjects X 1 dose
  MAD 1 placebo 2 subjects x 3 doses MAD 2 placebo 2 subjects x 3 doses MAD 3 placebo 2 subjects x 3 doses
  Interventions: Drug: JUV-161, Placebo

INTERVENTIONS:
Drug: JUV-161, Placebo — Single-Ascending, Placebo-Controlled

SUMMARY:
The present First-In-Human (FIH) study (JUV-161-101) aims to assess the safety, tolerability, and pharmacokinetics (PK) of single and multiple subcutaneous (SC) doses of JUV-161 in healthy volunteers. The study design is well-established for FIH studies and appropriate to assess the preliminary safety and tolerability of new drug candidates.

Data from this study will support conduct studies in patients with DM1 as well as supporting studies in other degenerative myopathies and other disorders for which preclinical efficacy data have been obtained.JUV-161 has not been previously been administered to human subjects.

DETAILED DESCRIPTION:
This is a FIH, randomized, double-blind, placebo-controlled, single- and multiple-ascending dose study. The study will be conducted at a single center and will include healthy volunteer subjects.

Enrollment in the SAD portion of the study will include up to 6 cohorts of 8 healthy adult volunteer subjects each of whom will receive a single dose of study drug (JUV-161, n=6; placebo, n=2). Enrollment in the MAD portion of the study will include up to 3 cohorts of 8 healthy adult volunteer subjects each of whom will receive multiple doses of study drug (JU161, n=6; placebo=2) For dosing, consideration of all relevant information obtained from in vitro and nonclinical toxicity studies was used to estimate no observed adverse effect levels (NOAELs) and a human equivalent dose (HED). Data from a 1-month non-human primate (cynomolgus monkeys) GLP study indicated that the NOAEL (HED) was ≥ 10 mg/kg. Using data from this study, modeling predicts that in humans the time to maximal concentration (Tmax) of JUV-161 will be 30-36 hours and the expected half-life (T1/2) of JUV-161 in humans will be approximately 80 hours.

Based on this information, the planned starting dose of JUV-161 0.10 mg/kg was selected to mitigate known, unknown or theoretical risks associated with administration of JUV-161. Sentinel dosing will be implemented within each SAD cohort as an additional safety measure to enable detection of possible acute safety risk(s).

In each SAD cohort, 2 subjects (1 JUV-161 and 1 placebo) will receive Study Drug on Study Day 1 (sentinel dosing). Following administration of study drug, a 72-hour period will be observed to detect the occurrence of reactions or significant adverse events (AEs). If safety and tolerability results are acceptable, 3 subjects will be dosed on Study Day 4. Following an additional 72-hour period and assuming no significant safety issues are identified, the final 3 subjects will be dosed on Study Day 7.

A Safety Review Committee (SRC) will conduct two Safety Reviews per SAD dosing Cohorts only.

On Study Day 3 of each SAD Cohort, the DMC SRC will review available clinical (including adverse events) and laboratory data from the Sentinel Dosing group to assess initial safety and tolerability of study drug. Assuming no safety issues are identified, dosing will proceed as described above.

On Study Days 28 through 35 of each Cohort, after completion of dosing for each subject in the Cohort, the SRC will review available clinical (including adverse events) and laboratory data to assess initial safety and tolerability of study drug. The review will include clinical, laboratory and (as available) pharmacokinetic data through 20 days after administration of Study Drug to the final 3 subjects in the Cohort. This period includes, and extends beyond, the predicted 5 half-lives of serum concentration following administration of JUV-161 for all subjects. Assuming no safety issues are identified, dosing for the subsequent Cohort may be initiated.

Additional study cohorts may be added, pending approval by the SRC, if the Sponsor believes additional dosing, safety, or pharmacokinetic data are required.

Enrollment in the MAD portion of the study will include at least 3 cohorts of 8 healthy adult volunteer subjects. Each subject will receive study drug (JUV-161, n=6; placebo, n=2) weekly X3 (Study Days 1, 8, 15). Additional study cohorts may be added, pending approval by the SRC, if the Sponsor believes additional dosing, safety, or pharmacokinetic data are required.

For the MAD cohorts, the dose range of 1.0 mg/kg to 5.0 mg/kg SC was chosen based on available safety data, a predicted efficacious dose for patients with DM1 (approximately 1 mg/kg SC once every week) and a practical SC dosing limitation.

Following successful review of safety data following dosing in SAD Cohorts 1 through 3, assuming no safety issues have been identified, Study Drug dosing for Cohort MAD 1 may begin.In each cohort, 8 subjects will receive study drug (JUV-161, n=6; placebo, n=2). At the discretion of the investigator and considering study site requirements, administration of study drug in the respective cohorts may occur on the same day (full cohort enrollment) or subjects may be broken into sub cohorts with administration of study drug on separate days (split cohort enrollment).At least 18 days following conclusion of dosing of the last subject in the Cohort, safety data will be reviewed by the SRC. As noted above, 18 days exceeds the predicted 5 half-lives following SC administration of JUV-161. SRC review will include available data for all subjects dosed in the Cohort (including clinical, laboratory, vital sign, ECG, and PK data and adverse event reports); these data will be assessed for safety and tolerability. Prior to SRC data review for MAD cohorts, at least 6 subjects will have received all 3 doses of Study Drug as described in the protocol. Assuming no safety issues are identified, dosing for the subsequent Cohort may be initiated. The safety review will be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Are males or nonpregnant females, ages 18 to 60 (inclusive) at time of signing Informed Consent with body mass index (BMI) 18 to 35 kg/m2
2. Are willing and able to give informed consent and follow all study procedures and requirements
3. Are able to understand the requirements of the study protocol
4. Agree to complete all required study visits
5. Are healthy, based on physical examination, medical history laboratory tests, vital signs and resting electrocardiograms
6. Are willing to abstain from caffeine and nicotine while in the Study Unit
7. Have negative screens for alcohol and drugs of abuse at screening and admission
8. Are willing to abstain from all alcoholic beverages and cannabinoids for 48 h prior to dosing through Post-dosing visit on Study Day 6.
9. Females must be either:

   * of non-childbearing potential (defined as having undergone surgical sterilization (hysterectomy, bilateral salpingectomy, bilateral oophorectomy or being postmenopausal (i.e., greater than 45 years old with amenorrhea for ≥ 12 months).) [Women under the age of 55 years must have a follicle stimulating hormone (FSH) level > 40mIU/mL to confirm menopause] OR
   * of child-bearing potential and using at least one of the following acceptable methods of contraception from at least 30 days prior to the time of informed consent through the time of study drug administration and for 8 weeks after last administration of study drug:

     1. Hormonal methods of contraception, including oral contraceptives containing combined estrogen and progesterone, a vaginal ring, injectable and implantable hormonal contraceptives, intrauterine hormone-releasing system (e.g., Mirena) and progestogen-only hormonal contraception associated with inhibition of ovulation
     2. Nonhormonal intrauterine device (IUD)
     3. Bilateral tubal occlusion
     4. Vasectomized subject/partner with documented azoospermia 90 days after procedure, if that partner is the sole sexual partner NOTE: WOCBP who are not exclusively in same-sex relationships must agree to use adequate contraception. WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, WOCBP must still undergo pregnancy testing as per protocol.

   NOTE: Complete abstinence, defined as the complete avoidance of heterosexual intercourse - is an acceptable form of contraception if used consistently throughout the duration of study and for the durations after dosing specified for males and females above. It is not necessary to use any other method of contraception when complete abstinence is elected. WOCBP who choose complete abstinence must continue to have pregnancy tests as per protocol. The reliability of sexual abstinence needs to be evaluated by the Investigator in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.

   NOTE: Female subjects must avoid egg donation from Screening through at least 2 months after administration of the last dose of study drug.
10. Men who are sexually active and males with partners of child-bearing potential must use the following forms of medically acceptable birth control during the study drug treatment period and for 16 weeks after the last administration of study drug:

    1. Vasectomy with medical assessment of surgical success and consistent use of a condom OR
    2. Consistent use of a condom with partner also using either stable hormonal contraceptive or IUD.

    NOTE: Males who are continuously not heterosexually active are exempt from contraceptive requirements.

    NOTE: Sperm donation is prohibited during the study and for up to 120 days4 months after the last administration of study drug.
11. Have NOT participated in a clinical study utilizing an investigational agent within 28 days or within 5 half-lives of the investigational drug (whichever is longer) prior to Screening

Exclusion Criteria:

1. Are unwilling or unable to comply with study procedures, including follow-up, as specified by the protocol, or unwilling to cooperate fully with the Investigator
2. Have a history of drug or alcohol abuse within 3 months of Screening
3. Have an active malignancy or have a history of malignancy within the 5 years prior to Screening. (Subjects with prior basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that were successfully treated may be enrolled.)
4. Have any of the following known active infections:

   1. Infection requiring systemic antiviral or antimicrobial therapy that would not have been completed within 30 days prior to screening
   2. Known history or positive test result for HIV, HBV or HCV
5. Have any clinical history or other active medical condition, psychiatric disorder or clinically significant laboratory abnormality, vital sign, ECG abnormality or other finding that, in the investigator's opinion, is likely to increase the risk of study participation, confound study results, or interfere with study conduct or adherence
6. Have any of the following:

   1. History of diabetes
   2. History of bleeding disorder or excessive bleeding
   3. Impaired renal function (estimated glomerular filtration rate [eGFR] <60ml/min/1.73m2, using the CKD-EPI (2021 equation) [See Appendix 1.]
   4. Platelet count < 125 X 109/L
   5. INR > ULN
   6. Electrocardiogram (ECG) showing QTcF > 470 msec female or > 450 msec male
7. Have received

   1. Treatment with any prescription medication within 14 days prior to screening (exception: contraceptives are permitted)
   2. Treatment with any non-prescription medication within 7 days or 5 half-lives (whichever is longer) prior to dosing (exception: acetaminophen up to 2 g per day prior to dosing is permitted)
   3. Any vaccination (therapeutic or prophylactic) within 30 days prior to screening and agree to not receive any vaccination during the course of the study
8. Prior exposure to JUV-161 or have known allergies to any components of the JUV-161 formulation
9. History of immune reaction to any biologic therapy
10. Donation or loss of greater than 1 unit (450 mL) of blood or donation of plasma through plasmapheresis within 7 days prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | From enrollment through to safety follow-up Visit on Day 60
Number of participants with treatment-emergent potentially clinically-significant safety abnormalities in safety laboratory parameters | From enrollment through to safety follow-up Visit on Day 60
Number of participants who have changes from baseline in electrocardiogram values in QTcF intervals | From enrollment through the safety follow-up visit on Day 60
Number of participants who have changes from baseline in heart rate ( beats per minute) | From enrollment through the safety follow-up visit on Day 60
Number of participants who have a change from baseline in systolic and diastolic blood pressure (mmHg) | From enrollment through the safety follow-up visit on Day 60

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Day 1 pre-dose and at 1, 2, 6, 12, 24, 36, 48, 60 and 72 hours Day 6,8,11,15,18,21 and 60
Time to the maximum measured plasma concentration (Tmax): | Up to 60 days
Area under the concentration-time curve from time zero through to infinity (AUC0-∞) | Up to 60 days.
Terminal elimination half-life in plasma (t1/2) | Up to 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Philip Ryan, MD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia